CLINICAL TRIAL: NCT03834402
Title: Interceptor Project: On Early Diagnosis Of The Prodromal Stage Of Alzheimer Disease. The Progression From Mild Cognitive Impairment (Mci) To Dementia: The Role Of Biomarkers In Early Interception Of Patients Candidate For Prescription Of Future Disease-Modifying Drugs
Brief Title: INTERCEPTOR Project: From MCI to Dementia
Acronym: INTERCEPTOR
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Ministry of Health, Italy (Other Government); Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Paolo Maria Rossini, Professor, Catholic University of the Sacred Heart
Other Study IDs: 2251
Record Dates: First submitted 2019-01-10; First posted 2019-02-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ApoE test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the next years a number of phase 2-3 trials which utilize experimental drugs possibly disease modifying for Alzheimer Dementia will reach their conclusion. This dense clinical trials activity has triggered a fundamental question both from Patients and Scientific Communities and Health Authorities/Insurances: on which basis will the new drugs -if effective-be distributed to patients or at-risk population? This question mainly deals with the "MCI prodromal to AD"condition since the MCI population actually includes about 50% of those who will progress to AD (the real "prodromic to AD" MCI form) while the remaining 50% will never convert to AD.

The INTERCEPTOR project is focused on the prodromic AD condition (IWG2) or the MCI condition (NIA-AA) which form the neuropsychological point of view and is characterized by means of: cognitive questionnaires, screening test (MMSE), extended neuropsychological evaluation.

The study is an observational, longitudinal cohort one, in which the baseline clinical and biomarkers characteristics of the enrolled MCI subjects at baseline will be compared for those classified as "AD converters" after 3.0 years of follow-up with respect to those "non-converters". MCI subjects who will convert to other forms of dementia will be examined separately. It will be considered the conversion to Alzheimer's disease within 3.0 years after diagnosis of MCI, together with the assessment of those who remain in a stable condition and those who have a reversion to normal cognitive profile. People with MCI who convert to other forms of dementia will be considered separately. The biomarker or a set of biomarkers that can predict the conversion to Alzheimer's disease with higher accuracy will be evaluated.

DETAILED DESCRIPTION:
In the next 8 years a number of phase 2-3 trials will end up which utilize experimental drugs possibly disease modifying for Alzheimer Dementia. They target different disease stages: mild-moderate AD, 'early' AD, MCI prodromic to AD (MCI + for biomarkers heralding progression to AD), pre-symptomatic AD in pathogenetic gene mutation carriers of familiar AD forms. This dense clinical trials activity has triggered a fundamental question both from Patients and Scientific Communities and Health Authorities/Insurances: on which basis will the new drugs -if effective-be distributed to patients or at-risk population? This question mainly deals with the "MCI prodromal to AD"condition since the MCI population actually includes about 50% of those who will progress to AD (the real "prodromic to AD" MCI form) while the remaining 50% will never convert to AD. Since the new drugs -if effective- will carry both elevated unit costs and not marginal side-effects, they should be administered selectively to those MCI with a severely high risk of conversion (i.e. 90% or more) and particularly to those with a highrisk of rapid conversion (1-2 years from diagnosis of the MCI condition).

The INTERCEPTOR project is focused on the prodromic AD condition (IWG2) or the MCI condition (NIA-AA) which form the neuropsychological point of view and is characterized by means of: cognitive questionnaire, screening test (MMSE), extended neuropsychological evaluation (incl. 2 episodic memory tests, language test, visuo-spatial abilities evaluation, behavioural scales, functional scales (Annex), full neurological examination. CDR must be 0.5. Atypical types of clinical presentations must be particularly considered (i.e. non amnesic debut) for a differential diagnosis where the role of biomarkers is pivotal.

In Italy, according to a recent study, an MCI prevalence of 5.9% has been evaluated in over 60 yrs population, with an increase of 4.5% between 60 & 69 yrs, of 5.8% between 70 & 79 yrs, and up to 7.1% in the 80 - 89 yrs range. On this epidemiological basis about 735.000 MCI cases are estimated for 2016in the resident Italian population. Multicentric non therapeutic cohort study in subjects fulfilling the MCI "core" criteria as defined by the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. The study design reflect a longitudinal cohort study in which the baseline clinical and biomarkers characteristics of the enrolled MCI subjects at baseline will be compared for those classified as "AD converters" after 3.0 years of follow-up with respect to those "non-converters". MCI subjects who will convert to other forms of dementia will be examined separately.

All the medications at baseline are allowed without modifications for the whole protocol except for urgencies.

Neuropsychological follow-up tests will be carried out at 6 months intervals (total 7 from T0= baseline to T6= 42 months).

Within 60 days from T0 biomarkers must be carried out/collected including:

MMSE & DRF - FCSRT) DNA extraction and ApoE typing Lumbar Puncture for Beta/Tau metabolites EEG for brain connectivity with graph theory MRI + hippocampal volumetry (18F)FDG-PET

ELIGIBILITY:
Inclusion Criteria:

1. age between 50 and 85 years;
2. age and education corrected Mini Mental State Examination score equal or superior to 24/30;
3. Clinical Dementia Rating (CDR) global score of 0.5;
4. concerns about cognitive modifications, expressed as subjective complaints by the subject, or by impression by a close acquaintance or an expert clinician;
5. defective performance with reference to age and education matched controls in one cognitive domain (memory, executive function, attention, language, visuospatial function): if repeated assessments are available, evidence of performance decline;
6. preserved functional autonomy: the subject remains fully independent, even if specific performances may be slower, less efficient than usual level, with occasional errors;
7. no dementia: the cognitive modifications do not significantly hamper social function or work activities.

Exclusion Criteria:

1. history of cerebrovascular disease (i.e. stroke episodes), alcohol abuse, severe medical disorders associated with cognitive impairment (organ failures, endocrine disorders, in particular thyroid disease and B12/folates deficiency); neuroimaging evidence of other potential causes of cognitive decline (e.g. subdural haematoma, malignancy etc.); chronic treatment with psychotropic drugs; women in reproductive age;
2. history of malignancy < 5 years;
3. contraindications for Magnetic Resonance Imaging (MRI): pacemaker; spinal stimulators; defibrillator; any other condition incompatible with MRI acquisition;
4. presence of spinal malformations or any other contraindications to lumbar puncture, according to the investigator's judgement;
5. HIV infection;
6. use of drugs potentially affecting cognitive function, according to the investigator's judgement;
7. subjects are not allowed to participate in any trial with experimental drug;

Exclusion criteria specific to lumbar puncture:

Patients who refuse to or cannot temporarily interrupt antiplatelet or anticoagulant therapy 14 days prior to sampling visit.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MCI subjects
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
MCI converting to AD | 3 years
  Percentage of enrolled patients that convert from MCI to Alzheimer's disease within 3.0 years.

SECONDARY OUTCOMES:
PREDICTING BIOMARKERS | 4.5 years
  Identify the biomarker or the set of biomarker that predict, using statistical techniques, in the most precise way the "conversion from MCI to AD" event.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Maria Rossini, Prof, Principal Investigator — Catholic University of Sacred Heart
Locations (1):
- Policlinico Agostino Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will only be at the disposal of the recruiting centers involved in the study

REFERENCES:
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Appollonio I, Leone M, Isella V, Piamarta F, Consoli T, Villa ML, Forapani E, Russo A, Nichelli P. The Frontal Assessment Battery (FAB): normative values in an Italian population sample. Neurol Sci. 2005 Jun;26(2):108-16. doi: 10.1007/s10072-005-0443-4. PMID 15995827
- [Background] Arevalo-Rodriguez I, Smailagic N, Roque I Figuls M, Ciapponi A, Sanchez-Perez E, Giannakou A, Pedraza OL, Bonfill Cosp X, Cullum S. Mini-Mental State Examination (MMSE) for the detection of Alzheimer's disease and other dementias in people with mild cognitive impairment (MCI). Cochrane Database Syst Rev. 2015 Mar 5;2015(3):CD010783. doi: 10.1002/14651858.CD010783.pub2. PMID 25740785
- [Derived] Lombardo FL, Lorenzini P, Mayer F, Massari M, Piscopo P, Bacigalupo I, Ancidoni A, Sciancalepore F, Locuratolo N, Remoli G, Salemme S, Cappa S, Perani D, Spadin P, Tagliavini F, Redolfi A, Cotelli M, Marra C, Caraglia N, Vecchio F, Miraglia F, Rossini PM, Vanacore N; INTERCEPTOR Network. Development of a prediction model of conversion to Alzheimer's disease in people with mild cognitive impairment: the statistical analysis plan of the INTERCEPTOR project. Diagn Progn Res. 2024 Jul 25;8(1):11. doi: 10.1186/s41512-024-00172-6. PMID 39049042